CLINICAL TRIAL: NCT06720142
Title: Clinical and Radiographic Outcomes of Patients Treated With Mg OSTEOCRETE
Brief Title: Mg OSTEOCRETE Post-Treatment Outcomes
Status: Recruiting | Type: Observational
Sponsor: Santiago Lozano-Calderon (Other)
Collaborators: Bone Solutions Inc (Unknown)
Responsible Party: Sponsor-Investigator, Santiago Lozano-Calderon, Attending Orthopaedic Surgeon/Assistant Professor, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2024P003397
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cancer of Bone; Trauma; Aseptic Loosening of Orthopaedic Hardware
Keywords: bone defect; bone substitute; osteocrete
MeSH Terms: conditions — Bone Neoplasms; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Bone void following bone tumor resection: Patients are being targeted because they have already agreed to receive OSTEOCRETE as part of standard clinical care. They will complete surveys, blood draws to test for magnesium levels, and low-dose CT scans at various post-operative timepoints.
  Interventions: Device: Mg OSTEOCRETE as a bone void filler
- Bone defect caused by aseptic loosening of orthopaedic implants: Patients are being targeted because they have already agreed to receive OSTEOCRETE as part of standard clinical care. They will complete surveys, blood draws to test for magnesium levels, and low-dose CT scans at various post-operative timepoints.
  Interventions: Device: Mg OSTEOCRETE as a bone void filler
- Bone defect caused by trauma-related condition: Patients are being targeted because they have already agreed to receive OSTEOCRETE as part of standard clinical care. They will complete surveys, blood draws to test for magnesium levels, and low-dose CT scans at various post-operative timepoints.
  Interventions: Device: Mg OSTEOCRETE as a bone void filler

INTERVENTIONS:
Device: Mg OSTEOCRETE as a bone void filler — Patients will be treated with Mg OSTEOCRETE as per standard clinical care to fill defects in bone left by bone tumor resection
  Groups: Bone void following bone tumor resection
Device: Mg OSTEOCRETE as a bone void filler — Patients will be treated with Mg OSTEOCRETE as per standard clinical care to fill defects in bone left by aseptic loosening of orthopaedic hardware
  Groups: Bone defect caused by aseptic loosening of orthopaedic implants
Device: Mg OSTEOCRETE as a bone void filler — Patients will be treated with Mg OSTEOCRETE as per standard clinical care to fill defects in bone left by trauma-related conditions
  Groups: Bone defect caused by trauma-related condition

SUMMARY:
Mg OSTEOCRETE is a bone substitute used to fill a defect in bone caused by excision of a tumor, orthopaedic hardware that has become loosened, or a trauma-related condition. The aim of this study is to determine the amount of time it takes for bone to heal after treatment with Mg OSTEOCRETE, and to better understand the efficacy of this treatment through clinical and patient-reported outcomes.

DETAILED DESCRIPTION:
Bone voids in the skeletal system can result from trauma, infection, surgery, or oncologic disease. If these voids are not treated, they may lead to issues such as pathological fractures, treatment or hardware failure, and recurrence of disease. Various methods exist for addressing bone voids, primarily through the use of grafting materials. Autograft-bone harvested from another part of the same patient and transplanted into the void-is considered the "gold standard" because they fulfill all three criteria of the "ideal" void filler: they are osteoconductive, osteoinductive, and osteogenic. However, their use can be limited by availability and potential donor site complications, with up to 39% of patients reporting pain at the donor site.

Due to concerns with traditional bone grafting methods, there is growing interest in alternative options. While allografts carry a risk of disease transmission and xenografts are prone to immune rejection, synthetic bone graft substitutes offer a promising alternative. These substitutes, made from materials like calcium sulfate or calcium phosphate, address many issues associated with autografts and allografts. With improved understanding of their performance post-implantation, ongoing advancements are being made. This Clinical Investigation Plan outlines an observational study to evaluate clinical and radiographic outcomes with a particular synthetic bone graft substitute (Mg OSTEOCRETE™; Alliant Biotech, LLC; Grand Rapids, MI).

Mg OSTEOCRETE™ is a moldable/injectable magnesium-based void filler that provides stability while also increasing cell proliferation. Use of Mg OSTEOCRETE™ has been shown to advance the rate of mineralization with a result of enhanced bone regeneration for multiple types of orthopedic applications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older on the day of surgery
* has received or will receive Mg OSTEOCRETE as a component of their treatment at this institution in accordance with Instructions for Use for the implanted product
* Mg OSTEOCRETE is indicated for one of the following reasons:

  1. as a bone void filler following bone tumor resection, or;
  2. as an augment for defects causing aseptic loosening of orthopaedic implants, or;
  3. to help substitute bone for trauma-related conditions

Exclusion Criteria:

* any contraindication as per Instructions for Use for Mg OSTEOCRETE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients who are 18 years or older and receive Mg OSTEOCRETE™ as bone void filler as a component of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time to complete bone remodeling | Pre-operatively through one year after surgery
  To determine the time to complete bone remodeling after injection of a magnesium-based bone graft substitute (Mg OSTEOCRETE™), as determined by Hounsfield Units on computed tomography (CT) scan.

SECONDARY OUTCOMES:
Survey of patient-reported outcomes and safety and efficacy of OSTEOCRETE | Pre-operatively through one year after surgery
  To collect safety and efficacy data regarding the performance of Mg OSTEOCRETE™. To longitudinally assess the patient-reported clinical outcomes after injection of a magnesium-based bone graft substitute (Mg OSTEOCRETE™).

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Lozano-Calderon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wu F, Wei J, Guo H, Chen F, Hong H, Liu C. Self-setting bioactive calcium-magnesium phosphate cement with high strength and degradability for bone regeneration. Acta Biomater. 2008 Nov;4(6):1873-84. doi: 10.1016/j.actbio.2008.06.020. Epub 2008 Jul 10. PMID 18662897
- [Background] Zhang Z., Yang Z., Chen Z., et al. A study on bone cement containing magnesium potassium phosphate for bone repair. Cogent Biol 2018;4(1):1487255. Doi: 10.1080/23312025.2018.1487255.
- [Background] Waselau M, Samii VF, Weisbrode SE, Litsky AS, Bertone AL. Effects of a magnesium adhesive cement on bone stability and healing following a metatarsal osteotomy in horses. Am J Vet Res. 2007 Apr;68(4):370-8. doi: 10.2460/ajvr.68.4.370. PMID 17397291
- [Background] Gulotta LV, Kovacevic D, Ying L, Ehteshami JR, Montgomery S, Rodeo SA. Augmentation of tendon-to-bone healing with a magnesium-based bone adhesive. Am J Sports Med. 2008 Jul;36(7):1290-7. doi: 10.1177/0363546508314396. Epub 2008 Mar 4. PMID 18319348
- [Background] Yoshizawa S, Brown A, Barchowsky A, Sfeir C. Magnesium ion stimulation of bone marrow stromal cells enhances osteogenic activity, simulating the effect of magnesium alloy degradation. Acta Biomater. 2014 Jun;10(6):2834-42. doi: 10.1016/j.actbio.2014.02.002. Epub 2014 Feb 7. PMID 24512978
- [Background] Diaz-Tocados JM, Herencia C, Martinez-Moreno JM, Montes de Oca A, Rodriguez-Ortiz ME, Vergara N, Blanco A, Steppan S, Almaden Y, Rodriguez M, Munoz-Castaneda JR. Magnesium Chloride promotes Osteogenesis through Notch signaling activation and expansion of Mesenchymal Stem Cells. Sci Rep. 2017 Aug 10;7(1):7839. doi: 10.1038/s41598-017-08379-y. PMID 28798480
- [Background] Pernaa K, Koski I, Mattila K, Gullichsen E, Heikkila J, Aho A, Lindfors N. Bioactive glass S53P4 and autograft bone in treatment of depressed tibial plateau fractures - a prospective randomized 11-year follow-up. J Long Term Eff Med Implants. 2011;21(2):139-48. doi: 10.1615/jlongtermeffmedimplants.v21.i2.40. PMID 22043972
- [Background] Russell TA, Leighton RK; Alpha-BSM Tibial Plateau Fracture Study Group. Comparison of autogenous bone graft and endothermic calcium phosphate cement for defect augmentation in tibial plateau fractures. A multicenter, prospective, randomized study. J Bone Joint Surg Am. 2008 Oct;90(10):2057-61. doi: 10.2106/JBJS.G.01191. PMID 18829901
- [Background] Heikkila JT, Kukkonen J, Aho AJ, Moisander S, Kyyronen T, Mattila K. Bioactive glass granules: a suitable bone substitute material in the operative treatment of depressed lateral tibial plateau fractures: a prospective, randomized 1 year follow-up study. J Mater Sci Mater Med. 2011 Apr;22(4):1073-80. doi: 10.1007/s10856-011-4272-0. Epub 2011 Mar 23. PMID 21431354
- [Background] Hofmann A, Gorbulev S, Guehring T, Schulz AP, Schupfner R, Raschke M, Huber-Wagner S, Rommens PM; CERTiFy Study Group. Autologous Iliac Bone Graft Compared with Biphasic Hydroxyapatite and Calcium Sulfate Cement for the Treatment of Bone Defects in Tibial Plateau Fractures: A Prospective, Randomized, Open-Label, Multicenter Study. J Bone Joint Surg Am. 2020 Feb 5;102(3):179-193. doi: 10.2106/JBJS.19.00680. PMID 31809394